CLINICAL TRIAL: NCT00304772
Title: A Randomized Comparative Study of Fluconazole Versus Micafungin for the Treatment of Candida Bloodstream Infection in Non-Neutropenic Patients
Brief Title: Fluconazole Versus Micafungin for Candida Bloodstream Infection in Non-Neutropenic Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Subjects were not recruited as intended.
Sponsor: Kyoto University (Other)
Collaborators: Pfizer (Industry); Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Takeshi Morimoto, Professor of Medicine, Kyoto University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JCRID0502
Record Dates: First submitted 2006-03-17; First posted 2006-03-20 (Estimated); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Candidiasis; Sepsis
Keywords: Candida; bloodstream infection; fluconazole; micafungin; randomized controlled trial
MeSH Terms: conditions — Candidiasis; Sepsis; Torulopsis | interventions — Fluconazole; Micafungin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Fluconazole
- 2 (Active Comparator)
  Interventions: Drug: Micafungin

INTERVENTIONS:
Drug: Fluconazole — 400mg/day
  Arms: 1
Drug: Micafungin — 150mg/day
  Arms: 2

SUMMARY:
The purpose of this study is to verify the equivalence in clinical efficacy of fluconazole and micafungin for the treatment of Candida bloodstream infection in non-neutropenic patients.

DETAILED DESCRIPTION:
Candida bloodstream infection occurs in patients with poor general conditions and has poor prognosis with attributable mortality of more than 30%. Clinical efficacy of fluconazole for the treatment of Candida bloodstream infection has been reported in clinical studies, since 1985 when it placed on the market. Fluconazole has established a position as the first-line drug up to date. However, possibly associated with the increased use of fluconazole, increased frequency of Candida species or strains with low susceptibility to fluconazole has been pointed out. Micafungin, an antifungal echinocandin with a different antifungal mechanism from fluconazole, has been reported to show good in vitro activity to various Candida species and strains with fluconazole resistance, and has comparative clinical efficacy with fluconazole for esophageal candidiasis, while it has relatively low in vitro activity to certain Candida species. There is no comparative study of fluconazole versus micafungin against Candida bloodstream infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients in whom Candida species have been isolated from blood culture.
* Patients accompanied by systemic infectious symptoms during the period from 24 hours (h) before collection of blood culture showing a positive result.
* Patients aged 20 years or older on the date of registration.
* Patients who have not received systemic administration of antifungal agents or who have started such administration within 48 h.
* Patients in whom a central venous (CV) catheter has been removed during the period from 24 h before collection of blood culture showing a positive result to registration, or a CV catheter can be removed within 72 h after registration.
* Patients with no verified undrainable abscess with a diameter of at least 3 cm, or impassable occlusive lesions, which are possibly attributable to Candida species.
* Patients from whom written informed consent to participate in this study has been obtained (or from their legally acceptable representatives).
* Patients who have adequate neutrophil count and hepatic/renal function in the blood test performed within 72 h before registration.

Exclusion Criteria:

* Patients with a history of adverse reactions associated with fluconazole or micafungin.
* Patients who have been treated with fluconazole or micafungin for at least 1 week within 12 weeks.
* Patients with a history of detection of fluconazole non-susceptible Candida species within 12 weeks.
* Patients in whom the neutrophil count is predicted to decrease to below 500/mL.
* Patients who are not treated with terfenadine, triazolam, cisapride, and ergotamine, which are contraindicated for concomitant use with fluconazole.
* Patients who are determined to be ineligible by the investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-08; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Treatment success (completion of protocol treatment within 12 weeks and recurrence-free survival at 4 weeks after the completion of protocol treatment) | 12 weeks and 4 weeks

SECONDARY OUTCOMES:
Safety | 12 weeks and 4 weeks
Duration of protocol treatment period in patients with treatment success | 12 weeks and 4 weeks
Overall survival at 4 and 12 weeks | 12 weeks and 4 weeks
Recurrence in patients who completed protocol treatment | 12 weeks and 4 weeks
Occurrence and deterioration of endophthalmitis during protocol treatment | 12 weeks and 4 weeks
Treatment success according to causative species, antifungal susceptibility profile, underlying condition | 12 weeks and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Satoshi Ichiyama, MD, PhD, Study Chair — Professor of Medicine, Department of Clinical Laboratory Medicine, Kyoto University Hospital; Shunji Takakura, MD, PhD, Principal Investigator — Instructor in Medicine, Department of Clinical Laboratory Medicine, Kyoto University Hospital
Locations (1):
- Department of Clinical Laboratory Medicine, Kyoto University Hospital, Kyoto, Japan